CLINICAL TRIAL: NCT05842304
Title: Personalized Brain Functional Sectors (pBFS)-Guided rTMS Intervention for Aphasia After Ischemic Stroke: a Multi-center, Randomized, Parallel Controlled Study
Brief Title: Individualized Precision rTMS for Language Recovery in Patients After Ischemic Stroke: a Multi-center RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changping Laboratory (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPSA0290
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-05

CONDITIONS: Stroke, Ischemic; Aphasia
MeSH Terms: conditions — Ischemic Stroke; Aphasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active cTBS group (Active Comparator): active cTBS combined with conventional rehabilitation therapy
  Interventions: Device: active cTBS
- sham cTBS group (Sham Comparator): Sham cTBS combined with conventional rehabilitation therapy
  Interventions: Device: sham cTBS

INTERVENTIONS:
Device: active cTBS — Each patient will receive three 600-pulse cTBS stimulations per day, parted by two 15-minute rest periods (a total of 1800 pulses daily), for 21 consecutive days (3 weeks).
  Arms: active cTBS group
Device: sham cTBS — Each patient will receive three 600-pulse sham cTBS stimulations per day, parted by two 15-minute rest periods (a total of 1800 pulses daily), for 21 consecutive days (3 weeks).
  Arms: sham cTBS group

SUMMARY:
The current multi-center study aims to evaluate the efficacy and safety of pBFS-guided rTMS Neuromodulation Treatment for the rehabilitation of language functions in ischemic stroke aphasic patients.

DETAILED DESCRIPTION:
Increasing evidence suggests that rTMS has been effective in treating various psychological and neurological diseases, including treating post-stroke symptoms. Using the personalized brain functional sectors (pBFS) technique, we could precisely identify individualized brain functional networks and the personalized language-related stimulation site based on the resting-state functional MRI data. The current study proposes to conduct a multi-center, double-blinded, randomized and parallel controlled design trial, to investigate the efficacy and safety of pBFS-guided personalized TMS intervention in post-stroke aphasic patients.

Subjects will be randomly assigned to the following two groups: active continuous TBS (cTBS) group, or a sham control group. The allocation ratio will be 2:1. Subjects will receive a 3-week treatment for 21 consecutive days. The stimulation procedure will be assisted with real-time neuronavigation to ensure its precision.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 35 and 75 years (including 35 and 75 years).
2. Meet the diagnostic criteria of acute ischemic stroke (using the 2019 American Heart Association/American Stroke Association Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke and the 2018 Chinese Society of Neurology Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke in China). All lesions should be in the left hemisphere, and the course of disease should be more than or equal to 2 months and less than or equal to 1 year .
3. Meet the diagnostic criteria for aphasia according to the Chinese version of the Western Aphasia Battery (WAB), with a WAB-aphasia quotient less than 93.8.
4. First onset, or with a history of stroke without apparent sequelae ( scored≤1 on modified Rankin Scale score (mRS) before the current stroke).
5. Normal functioning language abilities before the stroke, with Mandarin as their native language and an educational level higher than primary school (more than 6 years' education).
6. Understand the trial and be able to provide informed consent.

Exclusion Criteria:

1. Patients with comorbid severe dysarthria (NIHSS item 10 dysarthria ≥ 2).
2. Aphasia caused by other diseases such as brain tumor, Parkinson's syndrome, motor neuron disease, cerebral hemorrhage, traumatic brain injury, etc.
3. Patients with MRI scan and TMS treatment contraindications, such as claustrophobia, cardiac pacemaker, cochlear implant or other metallic foreign body and any electronic device implanted in the body.
4. History of epilepsy (having at least 2 uninduced seizures more than 24h apart, or a diagnosis of epilepsy syndrome, or having seizures within the past 12 months).
5. Patients with severe combined cardiac, pulmonary, hepatic, renal and other systemic diseases that cannot be controlled by conventional medication.
6. Patients with comorbid disorders of consciousness ( NIHSS 1(a)≥1).
7. Patients with combined malignant hypertension (sudden and significant increase in blood pressure, with increased systolic and diastolic blood pressure, often persisting above 200/130 mmHg)
8. Patients with co-malignant neoplasm.
9. Patients with a life expectancy of less than 1 year due to causes other than stroke.
10. Patients with combined deafness, visual impairment, or severe cognitive impairment to the extent that they are unable to cooperate with the test.
11. Patients with severe depression, anxiety, or diagnosed with other mental disorders to the extent that they are unable to cooperate with the trial.
12. History of TMS, transcranial electrical stimulation and other neuromodulation treatments in the past 3 months.
13. History of alcohol, drug, and/or other abuse.
14. Patients with other test abnormalities judged by the investigator to be unsuitable for the trial.
15. Women of childbearing age who are pregnant or preparing for pregnancy.
16. Patients who are participating in other clinical research trials.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2025-05-10 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Change in the Western Aphasia Battery scores | baseline, end of the 21-day therapy
  The first four subsets of the WAB (Spontaneous Speech, Auditory verbal comprehension, Repetition, Naming and word finding) will be used to evaluate the participants' language ability impairments. A Chinese adapted version of WAB will be used. The scores from all four subsets will be calculated into an Aphasia Quotient, lower scores indicate worse outcomes.

SECONDARY OUTCOMES:
Change in the Western Aphasia Battery scores | baseline, end of the 7-day therapy, end of the follow-up of 3 weeks
  The first four subsets of the WAB (Spontaneous Speech, Auditory verbal comprehension, Repetition, Naming and word finding) will be used to evaluate the participants' language ability impairments. A Chinese adapted version of WAB will be used. The scores from all four subsets will be calculated into an Aphasia Quotient, lower scores indicate worse outcomes.
National Institute of Health stroke scale | baseline, end of the 21-day therapy
  The 11-item National Institutes of Health Stroke Scale (NIHSS) will be used to evaluate participants' degree of neural deficits after stroke. Each item is associated with a specific ability, each scores between 0 to 4. The individual scores will be summed to calculate a participant's total NIHSS score. The total possible score is between 0 to 42, higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, Ph.D., Study Chair — Changping Laboratory
Locations (1):
- China Rehabilitation Research Center, Beijing, China